CLINICAL TRIAL: NCT06287398
Title: A Trial to Assess the Safety and Efficacy of Epcoritamab-containing Combination Salvage Therapy Followed by Autologous Stem Cell Transplantation and Epcoritamab Consolidation in Patients With Relapsed Large B-cell Lymphoma
Brief Title: Epcoritamab (Epcor)-Containing Combination Salvage Therapy Followed by ASCT & Epcor Consolidation in Patients With Relapsed LBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL38
Record Dates: First submitted 2024-02-07; First posted 2024-03-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; DLBCL, Nos Genetic Subtypes; High Grade B-Cell Lymphoma, Not Otherwise Specified; Follicular Large Cell Lymphoma, Relapsed; Follicular Large Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Epcoritamab Treatment (Experimental): Single arm study - All patients undergo same treatment with Epcoritamab for salvage and consolidation phases.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Epcoritamab (Epcor) is a bispecific antibody recognizing the T-cell antigen CD3 and the B-cell antigen CD20. Epcor is a supplied as a concentrate for solution for intended subcutaneous injection. The dose must be prepared by a qualified pharmacist using aseptic technique.
  Epcoritamab-Salvage treatment phase:
  2-3 cycles of R-DHAOx therapy (rituximab, dexamethasone, cytarabine, oxaliplatin), given every 21 days combined with Epcoritamab subcutaneous weekly dosing (priming 0.16mg Cycle 1 Day 1, intermediate 0.8mg cycle 1 day 8, full dose 48mg from cycle 1 day 15 onwards)
  Epcoritamab Consolidation phase:
  6 cycles (28 days each) of subcutaneous Epcoritamab, commencing between 6-12 weeks post ASCT.
  Epcoritamab dosing and timing for consolidation:
  * Cycle 1 Day 1: Priming (0.16mg) dose
  * Cycle 1 Day 8: intermediate (0.8mg) dose
  * Cycle 1 Day 15: full dose 48mg
  * Cycle 1 Day 22, Cycle 2-3 Days 1, 8, 15 and 22: 48mg
  * Cycles 4 to 6 - Days 1 and 15 (fortnightly dosing): 48mg

SUMMARY:
The goal of this clinical trial is to evaluate clinical efficacy of incorporating Epcoritamab into the salvage treatment routine for relapsed-refractory aggressive B-cell lymphoma, followed by autologous stem-cell transplantation (ASCT) and consolidation Epcoritamab. The main questions it aims to answer are:

* Will the addition of epcoritamab to intensive salvage chemotherapy be safe and increase the proportion of patients with relapsed or refractory (R/R) large B-cell lymphoma who achieve a complete remission prior to planned transplant?
* Is consolidation epcoritamab after ASCT deliverable and safe?
* Will consolidation epcoritamab will result in improved clearance of molecularly detectable residual disease?
* Will the combination of pre- and post-ASCT epcoritamab lead to higher rates of progression-free survival (PFS) and event free survival (EFS) at 12 months compared to historical estimates in this population.

Participants will undergo three phases in this trial:

1. Epcoritamab-Salvage treatment: consists of 3 cycles of R-DHAOx (rituximab, dexamethasone, cytarabine, oxaliplatin) plus Epcoritamab
2. ASCT: Pre-autograft eligibility assessment for ASCT will be performed according to local practice. ASCT may be administered at local referring centre and will follow local standard operative procedures.
3. Consolidation treatment: consists of six 28-day cycles of subcutaneous Epcoritamab, commencing 6 - 12 weeks post ASCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Confirmed diagnosis of DLBCL, Not-otherwise specified (NOS), Transformation of indolent B-cell lymphoma, High-grade B-cell lymphoma (HGBCL), NOS, Diffuse-large BCL (DLBCL)/ High-grade B-cell lymphoma (HGBL) with MYC and BCL2 rearrangements or Follicular large B-cell lymphoma according to World Health Organization (WHO) 2016 or 2022 criteria that has relapsed or progressed after one line of chemoimmunotherapy
3. Transplant eligible according to local assessment
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Measurable disease on computed tomography (CT) scan, defined as a nodal site greater than 1.5cm in longest axis or an extranodal site greater than 1.0cm in longest axis AND baseline fluorodeoxyglucose (FDG) positron emission tomography (PET) scans must demonstrate positive lesion compatible with CT defined anatomical tumour sites
6. Histological confirmation of tumour CD20 positivity, analysed by immunohistochemistry, on a pre-enrolment tissue sample performed after most recent prior therapy
7. Adequate renal function

   - Creatinine clearance greater than 45mL per min (Cockcroft Gault formula)
8. Adequate hepatic function:

   * Aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 3x Upper Limit of Normal (ULN)
   * Bilirubin less than or equal to 1.5x Upper Limit of Normal (ULN) or less than or equal to 3 if documented liver involvement and/or Gilbert's disease.
9. Adequate haematologic function:

   * Haemoglobin greater than or equal to 90g/L (transfusion support permitted)
   * Absolute neutrophil count greater than or equal to 1.0 x 109 per L; growth factor support allowed in case of bone marrow involvement
   * Platelet count greater than 75 x 109 per L or greater than or equal to 50 x 109 per L if documented marrow involvement
10. Able to take oral medications
11. Adequate washout of prior therapies:

    * At least 4 weeks since last dose of immunochemotherapy, radio-conjugated or toxin-conjugated compound, or other investigational anti-cancer therapy
    * At least 6 weeks since chimeric antigen-receptor T-cell therapy
12. Resolution of toxicities from prior therapy to a grade that does not contraindicate trial participation in the opinion of the investigator
13. If receiving glucocorticoid treatment at screening, treatment must be tapered down and administered with a maximum of 25 mg daily in the last 14 days before the first dose of Epcoritamab
14. Before the first dose of Epcoritamab, during the trial and for 12 months after last administration of Epcoritamab, a woman must be either:

    1. Not of childbearing potential, defined as: premenarchal; postmenopausal (greater than 45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level greater than 40 IU per L or milli-International unit (mIU) per mL); permanently sterilized (e.g., bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
    2. Of childbearing potential and practicing a highly effective method of birth control (as defined by the European Clinical Trial Facilitation Group) consistent with local regulations regarding the use of birth control methods for patients participating in clinical trials: e.g., established use of oral, injected or implanted combined (estradiol and progesterone containing) hormonal contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); male partner sterilization (the vasectomized partner should be the sole partner for that patient); true abstinence (when this is in line with the preferred and usual lifestyle of the patient) * If the childbearing potential changes after start of the trial (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) a woman must begin a highly effective method of birth control, as described under 16b
15. A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control (that is the use of condom) during the trial and for 12 months after receiving the last dose of Epcoritamab
16. Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the trial and for 12 months after receiving the last dose of Epcoritamab. Men must also not donate sperm during the trial and for 12 months after receiving the last dose of Epcoritamab
17. The patient understands the purpose of the trial and procedures required for the trial and is capable of giving signed informed consent which includes compliance with the requirements (no medical or psychiatric reason precluding participation) and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Diagnosis of primary Central Nervous System (CNS) lymphoma
2. Active secondary CNS involvement of lymphoma at time of screening

   - A prior history of secondary CNS lymphoma is allowed provided that it has been successfully treated and there are no features of recurrence.
3. Prior autologous stem cell transplant
4. Known past or current malignancy other than inclusion diagnosis, except for:

   1. Cervical carcinoma of Stage 1B or less.
   2. Non-invasive basal cell or squamous cell skin carcinoma.
   3. Non-invasive, superficial bladder cancer.
   4. Prostate cancer with a current Prostate Specific Agent (PSA) level less than 0.1 ng per mL e. indolent lymphoma
   5. Indolent lymphoma
   6. Other malignancy that has been treated with curative intent and has remained in remission for 2 years
5. Any prior therapy with a bispecific antibody targeting CD3 and CD20
6. Uncontrolled systemic infection
7. Known HIV infection
8. Known active hepatitis B or C infection based on criteria below:

   * Hepatitis B virus (HBV): Patients with positive HbsAg are excluded. Patients with positive hepatitis B core antibody (antiHBc) and negative HbsAg require negative hepatitis B polymerase chain reaction (PCR) before enrolment and must be treated with antiviral therapy. Patients who are hepatitis B PCR positive will be excluded.
   * Hepatitis C virus (HCV): If positive hepatitis C antibody, patient will need to have a negative hepatitis C ribonucleic acid (RNA) before enrolment. Patients who are hepatitis C RNA positive will be excluded.
9. Seizure disorder, unless seizure-free for 12 months on established anticonvulsant therapy without the requirement for modification to anticonvulsants within the prior 12 months
10. Known clinically significant cardiac disease, including:

    1. Onset of unstable angina pectoris within 6 months of signing the patient informed consent form (PICF)
    2. Acute myocardial infarction within 6 months of signing the PICF
    3. Congestive heart failure (grade III or IV as classified by the New York Heart Association
    4. Decreased ejection fraction of less than 45%
11. Confirmed history or current autoimmune disease requiring permanent immunosuppressive therapy. Low-dose prednisolone (less than or equal to 10mg/day or equivalent) for rheumatoid arthritis or similar conditions is allowed.
12. Exposed to live or live attenuated vaccine within 4 weeks prior to signing PICF
13. Women who are pregnant or lactating.
14. Patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
15. Known hypersensitivity or adverse reaction to rituximab, tocilizumab or any elements of DHAOx
16. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. This condition must be discussed with the patient prior to signing consent and registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 12 months
  Time to event outcome measured in days from commencement of each treatment subset (salvage chemotherapy and Epcoritamab/ASCT/ Epcoritamab re-treatment) to date of first to occur out of reduced partial response (PR) after C2, commencement of non-protocolised cancer treatment, progression or death from any cause.

SECONDARY OUTCOMES:
Evaluate safety and tolerability of combination Epcoritamab with salvage-ASCT | From enrolment to 30 days after the final treatment is completed.
  Rate of adverse events according to CTCAE criteria v 6.0 expressed as a number and proportion.
Overall response rate (ORR) | At cycle 2 day 21 (each cycle is 28 days), cycle 3 day 21, 4 weeks post ASCT, 12 months from registration and 3-monthly during follow up (up to 24 months from registration).
  Defined as achievement of at least a partial response to treatment according to Lugano criteria i.e. achievement of a PR or CR at any time during study participation
Complete response rate (CRR) | At cycle 2 day 21 (each cycle is 28 days), cycle 3 day 21, 4 weeks post ASCT, 12 months from registration and 3-monthly during follow up (up to 24 months from registration).
  Defined as achievement of CR at any time during study according to Lugano criteria
Overall Survival (OS) | At cycle 2 day 21 (each cycle is 28 days), cycle 3 day 21, 4 weeks post ASCT, 12 months from registration and 3-monthly during follow up (up to 24 months from registration).
  Defined as the time from commencement of study treatment until death from any cause
Progression free survival (PFS) | At cycle 2 day 21 (each cycle is 28 days), cycle 3 day 21, 4 weeks post ASCT, 12 months from registration and 3-monthly during follow up (up to 24 months from registration).
  Defined as the time from commencement of study treatment until disease progression or death from any cause, following Epcoritamab-chemotherapy salvage, transplant and maintenance. Time to event outcome measured in months.

CONTACTS AND LOCATIONS:
Locations (1):
- Australasian Leukemia and Lymphoma Group, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared publicly. Aggregate patient data and final results will be presented in the final report.